CLINICAL TRIAL: NCT00332007
Title: A Single Centre, Double-blind, Randomised, Placebo Controlled Crossover Study to Evaluate the Efficacy and Tolerability of Tonabersat in the Prophylaxis of Migraine in Patients Presenting With Migraine With Aura
Brief Title: Tonabersat in the Prophylaxis of Migraine With Aura
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Minster Research Ltd (Industry)
Collaborators: University of Copenhagen (Other)
Responsible Party: Professor J Olesen, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: TON/02/05-CLIN
Record Dates: First submitted 2006-05-30; First posted 2006-05-31 (Estimated); Last update posted 2009-08-31 (Estimated); Status verified 2009-08

CONDITIONS: Migraine With Aura
MeSH Terms: conditions — Migraine with Aura | interventions — tonabersat

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Tonabersat 40 mg daily
  Interventions: Drug: Tonabersat
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tonabersat — two tablets once daily
  Arms: 1
Drug: Placebo — two tablets once daily
  Arms: 2

SUMMARY:
Overall trial objectives:

1. Can treatment with tonabersat reduce the number of days with aura and/or migraine headache in patients with migraine with aura
2. How well tolerated is treatment with tonabersat

The study is based on the hypothesis that the unique mechanism of action of tonabersat will inhibit some of the early events in the generation of aura and migraine headache and so be effective as prophylactic treatment

ELIGIBILITY:
Inclusion Criteria:

* Patients with an established history of migraine of at least one year meeting the diagnostic criteria of the International Classification of Headache Disorders - Edition 2 (Appendix 2) and who experience at least one aura a month.
* Male or female patients between 18-65 years of age
* Women of child bearing potential must be using a reliable form of contraception (defined in the protocol) for at least 3 months prior to enrolment and they must have a negative pregnancy test at screening with no intention of becoming pregnant during the study period

Exclusion Criteria:

* Patients experiencing headache other than migraine or tension headache
* Overuse of acute migraine treatments defined as more than 14 daily doses per month with analgesics or more than 9 daily doses per month of ergots or triptans within the last two months
* Migraine prophylactic treatment within two months prior to entry to the trial
* Patients taking any of the following medications for migraine: beta-blockers, tricyclic antidepressants (during the last 2 months), antiepileptic dugs (during the last 2 months), calcium channel blockers, monoamine oxidase inhibitors, daily NSAIDs, daily paracetamol, high dose magnesium supplements (600mg/day). Parenteral administration of botulinum toxin is also excluded. These drugs are permitted when given for diseases other than migraine provided that, in the opinion of the investigator the dose can be kept constant throughout the trial.
* Patients who, in the opinion of the investigator, have significant cerebrovascular disease e.g. transient ischaemic attacks, stroke
* Patients who, in the opinion of the investigator, have clinically significant cardiovascular disease
* Patients suffering from a current clinical diagnosis of a major depressive disorder or schizophrenia
* Patients with renal dysfunction , defined as a serum creatinine of greater than 125% of the upper limit of normal for their age group
* Patients with hepatic dysfunction defined as a liver function test (AST, ALT, alkaline phosphatase, bilirubin) of greater than twice the upper limit of normal for their age group
* Patients with known alcohol or other substance abuse
* Use of an investigational drug (for any indication) within 30 days or 5 half-lives, whichever is the longer, prior to screening
* Women who are pregnant or breast feeding
* Women of childbearing potential not using a reliable form of contraception
* Patients with any other clinically significant condition which, in the investigators opinion, would render them unsuitable for this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2006-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Difference in the mean number of aura attacks experienced between treatment groups | 12 week treatment period
Difference in the mean number of migraine headache days between treatment groups | 12 week treatment period
Incidence of adverse events | 12 week treatment period

SECONDARY OUTCOMES:
Mean number of headache days in each treatment period. | 12 week treatment period
Mean number of auras followed by headache in each treatment period. | 12 week treatment period
Mean number of headache days in each month of treatment in each treatment period. | Mean monthly
Mean number of auras and/or migraine headache during each treatment period. | 12 week treatment period
Mean number of migraine headache attacks in each treatment period. | 12 week treatment period
Speed of effect of treatment. | First month for which difference between treatments identified
Mean monthly consumption of rescue medication. | Mean monthly
Mean duration of auras in each treatment period. | Mean over 12 week treatment period
Mean number of symptoms associated with auras in each treatment period. | 12 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Jes Olesen, MD, Principal Investigator — University of Copenhagen, Department of Neurology, Glostrup Hospital
Locations (1):
- Danish Headache Centre, Department of Neurology, Glostrup Hospital, Copenhagen, Denmark

REFERENCES:
- [Background] International Headache Society Clinical Trials Subcommittee. Guidelines for controlled trials of drugs in migraine (second edition). Cephalalgia 2000; 20:765-86. Committee for Proprietary Medicinal Products. Note for guidance on clinical investigation of medicinal products for the treatment of migraine, CPMP/EWP/788/01/Final. London, 17 December 2003.
- [Background] Committee for Proprietary Medicinal Products. Note for guidance on clinical investigation of medicinal products for the treatment of migraine, CPMP/EWP/788/01/Final. London, 17 December 2003.
- [Result] Hauge AW, Asghar MS, Schytz HW, Christensen K, Olesen J. Effects of tonabersat on migraine with aura: a randomised, double-blind, placebo-controlled crossover study. Lancet Neurol. 2009 Aug;8(8):718-23. doi: 10.1016/S1474-4422(09)70135-8. Epub 2009 Jun 29. PMID 19570717